CLINICAL TRIAL: NCT01248247
Title: BATTLE-2 Program: A Biomarker-Integrated Targeted Therapy Study in Previously Treated Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH); GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0360; P01 CA148133 (Other Grant/Funding Number: NCI); NCI-2011-01104 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Lung Cancer
Keywords: Non small cell lung cancer; Biopsy accessible tumor; Stage IIIB non small cell lung cancer; Stage IV non small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; AZD 6244; MK 2206; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 - Erlotinib (Experimental): Erlotinib 150 mg by mouth each day of a 28 day cycle.
  Interventions: Drug: Erlotinib
- Group 2 - Erlotinib + MK-2206 (Experimental): Erlotinib 150 mg by mouth each day of a 28 day cycle.
  MK-2206 135 mg by mouth every week of a 28 day cycle.
  Interventions: Drug: Erlotinib; Drug: MK-2206
- Group 3 - AZD6244 + MK-2206 (Experimental): AZD6244 100 mg by mouth daily of a 28 day cycle. MK-2206 100 mg by mouth every week of a 28 day cycle.
  Interventions: Drug: AZD6244; Drug: MK-2206
- Group 4 - Sorafenib (Experimental): Sorafenib 400 mg by mouth twice a day for a 28 day cycle.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Erlotinib — 150 mg by mouth each day of a 28 day cycle.
  Other Names: OSI-774; Tarceva
  Arms: Group 1 - Erlotinib
Drug: AZD6244 — 100 mg by mouth daily of a 28 day cycle.
  Arms: Group 3 - AZD6244 + MK-2206
Drug: MK-2206 — 100 mg by mouth every week of a 28 day cycle.
  Arms: Group 3 - AZD6244 + MK-2206
Drug: Sorafenib — 400 mg by mouth twice a day for a 28 day cycle.
  Other Names: Nexavar; BAY43-9006
  Arms: Group 4 - Sorafenib
Drug: Erlotinib — 150 mg by mouth daily of a 28 day cycle.
  Other Names: OSI-774; Tarceva
  Arms: Group 2 - Erlotinib + MK-2206
Drug: MK-2206 — 135 mg by mouth every week of a 28 day cycle.
  Arms: Group 2 - Erlotinib + MK-2206

SUMMARY:
Different people have different biomarkers (chemical "markers" in the blood that may be related to your reaction to study drugs). If researchers know about your biomarkers before you receive treatment, they may be able to prescribe a treatment that is better suited to your body's specific needs.

The goal of this clinical research study is to learn if drug or drug combinations based on your biomarkers can help to control NSCLC. The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Erlotinib hydrochloride, MK-2206, AZD6244, and Sorafenib are targeted therapies. Targeted therapy is a type of drug that blocks the growth of cancer cells by interfering with specific targeted molecules needed for tumor growth, rather than by simply interfering with rapidly dividing cells (for example with traditional chemotherapy).

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 4 groups:

* If you are in Group 1, you will take erlotinib alone.
* If you are in Group 2, you will take erlotinib and MK-2206.
* If you are in Group 3, you will take AZD6244 and MK-2206.
* If you are in Group 4, you will take sorafenib alone.

The group you are in will be assigned by a computer. The results of your screening tests will be used to determine (and may limit) which of the 4 groups you may be eligible to be assigned to. Your likelihood of being in any 1 group over another may also be affected by how well that treatment has done in earlier study participants. Your study doctor will tell you which group you have been assigned.

Study Drug Administration:

Each cycle is 28 days.

* If you are in Group 1, you will take erlotinib hydrochloride by mouth 1 time every day.
* If you are in Group 2, you will take MK-2206 by mouth 1 time every week. You will take erlotinib hydrochloride by mouth 1 time every day.
* If you are in Group 3, you will take MK-2206 by mouth 1 time per week. You will take AZD6244 by mouth 1 time every day.
* If you are in Group 4, you will take sorafenib by mouth 2 times every day.

If you will take erlotinib hydrochloride (Groups 1 and 2), you should take the tablets in the morning. You should take the drug 1 hour before or 2 hours after a meal, with no more than 7 ounces of water. If you forget to take a dose, the last missed dose should be taken as soon as you remember, as long as it is at least 12 hours before the next dose. The next day, you should take the scheduled dose at the usual time. You should try not to vomit for at least 30 minutes after taking the drug. If you feel nauseated before or after taking the erlotinib, you should take an anti-nausea drug. You may take an extra dose of erlotinib if you vomit within 30 minutes after taking the tablet.

If you are in Group 2, you should take MK-2206 at about the same time each week with about 1 cup (8 ounces) of water. You must take MK-2206 at least 2 hours before or at least 2 hours after any food or a meal. You should not make up any missed doses.

If you are in Group 3, you should take MK-2206 at about the same time each week with about 1 cup (8 ounces) of water. You must take MK-2206 at least 2 hours before or at least 2 hours after eating. You should not make up any missed doses.

If you will take AZD6244 (Group 3), you should take the study drug in the morning before you eat or drink anything. You can eat breakfast 1 hour after you take the dose.

If you will take sorafenib, you must take your doses 12 hours apart. You will take 2 tablets each morning, and again each evening. Sorafenib should be taken with about 1 cup of water on an empty stomach (either 1 hour before a meal or 2 hours after a meal). If you feel nauseated before or after taking the medication, anti-nausea medications should be used. If you miss a dose, you should skip it and take the next scheduled dose at the right time.

Your medication should be stored at room temperature.

Study Visits:

The study visit schedule is described below. In certain cases, with the permission of your doctor, the study visits may occur up to 7 days earlier or later than described below.

On Day 1 of each cycle:

* You will have a complete physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests. If your doctor thinks it is needed, you may have to have these blood tests more often.

On Day 1 of every odd-numbered cycle (Cycles 3, 5, 7, and so on):

* You will have a CT scan and/or MRI of the chest (and abdomen if the doctor thinks it is needed) to check the status of the disease.
* You will have a chest x-ray.
* MRI of the brain (if the doctor thinks it is needed)

Additional Tests for Group 2:

* During screening, on Day 1 of Cycle 2, and at the end-of study visit, you will have an eye exam.
* On Day 1 of Cycle 1 you will have an ECG before taking your study medication and then again about 4 hours after you take your study medication.

Additional Tests for Group 3:

* During screening, on Day 1 of Cycle 2, and at the end-of study visit, you will have an eye exam.
* During Cycle 2 (Week 6 of being on study drug), on Day 1 of Cycle 4, and then every 3 months, you will have a multigated acquisition (MUGA) scan and/or echocardiogram to check your heart function. You will have these tests more often if the doctor thinks it is needed.
* On Day 1 of Cycle 1 you will have an ECG before taking your study medication and then again about 4 hours after you take your study medication.

Length of Study:

You may continue to take the study drug(s) for as long as you are benefitting. You will be taken off study if the disease gets worse or if you have intolerable side effects.

End-of-Study Visit:

When you go off study for any reason, you will have an end-of-study. This visit may occur up to 7 days earlier or later. The following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a complete physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) and urine will be collected for routine tests.
* You will have a CT scan and/or MRI of the chest (and abdomen if the doctor thinks it is needed) to check the status of the disease.
* You will have a chest x-ray.
* You will have an ECG (Group 3).

Follow-Up:

You will have a follow-up evaluation performed 4 weeks ± 7 days after therapy is discontinued. This evaluation may be a visit or contact by phone by the research personnel. If you are in Group 3, you will have a MUGA scan and/or echocardiogram to check your heart function.

You will be called every 3 months for up to 3 years and asked about any cancer treatments you may be receiving. This phone call will take about 10 minutes.

This is an investigational study. Erlotinib is FDA approved and commercially available for treatment of NSCLC that has gotten worse. Sorafenib is approved in renal cell cancer and hepatocellular carcinoma. Sorafenib has also has also been evaluated in unselected advanced patients with NSCLC both alone or with chemotherapy in the first-time treatment of patients . MK-2206, and AZD6244 are not FDA-approved or commercially available. At this time, they are only being used in research.

Up to 450 patients will take part in this multicenter study. Approximately 350 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a diagnosis of pathologically confirmed NSCLC by tumor biopsy and/or fine-needle aspiration.
2. The subject has a diagnosis of either advanced, incurable stage IIIB or stage IV NSCLC, and failed at least one front-line metastatic NSCLC chemotherapy regimen, or EGFR TKI. (Subjects who have failed adjuvant or locally advanced therapy within 6 months are also eligible to participate in the study).
3. The subject has measurable NSCLC (patients with active new disease growth in previously irradiated site are eligible).
4. The subject's ECOG performance status is </= 2 at study entry.
5. The subject has biopsy accessible tumor
6. The subject has adequate hematologic function as defined by an absolute neutrophil count (ANC) >/= 1,500/mm3, platelet count >/= 100,000/mm3, WBC >/= 3,000/ mm3, and hemoglobin >/= 9 g/dL.
7. The subject has adequate hepatic function as defined by a total bilirubin level </= 1.5 x the upper limit of normal (ULN) (bilirubin >/= 1.5 x ULN with known Gilbert's disease is allowed), and alkaline phosphatase, AST and ALT </= 2.5 x the upper limit of normal or </= 5.0 x ULN if liver metastases are present.
8. Serum creatinine clearance >50ml/min, either by Cockcroft-Gault formula or 24-hour urine collection analysis
9. If subject has brain metastasis, they must have been stable (treated and/or asymptomatic) and off steroids for at least 2 weeks.
10. The subject is >/=18 years of age.
11. The subject has signed informed consent.
12. The subject is eligible if disease free from a previously treated malignancy, other than a previous NSCLC, for greater than two years. Subject with a history of prior basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix are allowed.
13. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Childbearing potential will be defined as women who have had menses within the past 12 months, who have not had tubal ligation, hysterectomy or bilateral oophorectomy. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately.
14. The subject, if a man, agrees to use effective contraception or abstinence while on study and for 90 days after last dose of study drug.
15. Subject is able to swallow capsules and has no surgical or anatomical condition that will preclude the patient from swallowing and absorbing oral medications on an ongoing basis.

Exclusion Criteria:

1. The subject has received prior chemotherapy, surgery, or radiotherapy within 3 weeks of initiating study drug, or 4 weeks for bevacizumab or investigational drug or 72 hours for erlotinib or the subject has not recovered (</= Grade 1) from side effects of the prior therapy (localized palliative radiotherapy within 2 weeks is allowed).
2. The subject has undergone prior thoracic or abdominal surgery within 30 days of study entry, excluding prior diagnostic biopsy.
3. The subject has cardiac conditions as follows: uncontrolled hypertension BP > 140/90 despite optimal therapy, uncontrolled angina, ventricular arrhythmias, or congestive heart failure New York Heart Association Class II or above, baseline LVEF </= 50%, prior or current cardiomyopathy, atrial fibrillation with heart rate >100 bpm, unstable ischaemic heart disease (MI within 6 months prior to starting treatment, or angina requiring use of nitrates more than once weekly).
4. The subject has neuropathy >/= grade 2
5. The subject is pregnant (confirmed by serum b-HCG if applicable) or is breastfeeding. In the event of inconclusive pregnancy test results, the investigator will have final determination of pregnancy status.
6. Subjects will be excluded for other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, severe infection requiring active treatment, severe malnutrition, chronic severe liver or renal disease).
7. Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
8. Subjects with poorly controlled diabetes (HbA1c >8%) are excluded.
9. Subjects whose tumor harbors the EML4-ALK fusion gene are excluded unless the patient has failed treatment with Anaplastic Lymphoma Kinase (ALK) inhibitor.
10. Subjects are excluded if they have QTc prolongation >450 msec (Bazett's Formula) for males or >470 ms for females on screening or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) including heart failure that meets New York Heart Association (NYHA) class II or above or require use of a concomitant medication that can prolong the QT interval.
11. Subjects who have abnormal K+ or Mg++ levels will be excluded if these levels cannot be corrected to within normal range with adequate supportive treatment prior to study drug initiation.
12. Subjects whose tumor harbors an EGFR mutation are excluded unless the subject failed treatment with EGFR TKIs in which case the subject can be randomized to Arms 2, 3, and 4.
13. Drug Specific Eligibility Criteria based on Treatment Arms- Subjects are excluded from the erlotinib monotherapy arm if they have progressed on prior EGFR TKI therapy; from the AKT inhibitor arm(s) if they have received prior AKT inhibitor therapy; from the MEK inhibitor arm if they have received prior MEK inhibitor therapy; and from Sorafenib arm if they have previously received the drug or have prior history of clinically significant hemoptysis or bleeding diathesis as per principal investigator judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2011-06-02 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo V. Negrao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Yale Universtiy, New Haven, Connecticut
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with pretreated NSCLC who agreed to a baseline tumor biopsy, who had ECOG P of 0 to 2, and who had multiple prior lines of therapy and stable or treated brain metastases were enrolled. Patients were excluded if their tumor harbored EGFR sensitizing mutations or ALK gene fusions, and they were erlotinib or crizotinib na¨ıve.
Pre-assignment Details: Total of 334 participants consented, 134 participants did not receive treatment a majority due to screen failures and others due to participants withdrew consent(s) and or progressed prior to treatment starting.
Groups:
- Arm 1 - Erlotinib: Erlotinib 150 mg by mouth each day of a 28 day cycle.
- Arm 2 - Erlotinib + MK-2206: Erlotinib 150 mg by mouth each day of a 28 day cycle. MK-2206 135 mg by mouth every week of a 28 day cycle.
- Arm 3 - AZD6244 + MK-2206: AZD6244 100 mg by mouth daily of a 28 day cycle. MK-2206 100 mg by mouth every week of a 28 day cycle.
- Arm 4 - Sorafenib: Sorafenib 400 mg by mouth twice a day for a 28 day cycle.
Period: Overall Study
Arm/Group | Arm 1 - Erlotinib | Arm 2 - Erlotinib + MK-2206 | Arm 3 - AZD6244 + MK-2206 | Arm 4 - Sorafenib
Started | 22 | 42 | 75 | 61
Completed | 0 | 0 | 0 | 0
Not Completed | 22 | 42 | 75 | 61
Not completed — Adverse Event | 2 | 4 | 4 | 2
Not completed — Death | 0 | 1 | 4 | 7
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Alternative treatment | 0 | 1 | 0 | 0
Not completed — Other | 2 | 8 | 8 | 5
Not completed — Progression | 18 | 27 | 56 | 44
Not completed — Refuse further treatment | 0 | 0 | 1 | 2
Not completed — Complicating disease | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Erlotinib | Arm 2 - Erlotinib + MK-2206 | Arm 3 - AZD6244 + MK-2206 | Arm 4 - Sorafenib | Total
Number analyzed (Participants) | 22 | 42 | 75 | 61 | 200
Age, Continuous [Median (Full Range); unit: years] | 61 [34 to 82] | 62 [43 to 78] | 61 [26 to 76] | 62 [35 to 79] | 61 [26 to 82]
Age, Customized [Count of Participants; unit: Participants]
  <=49 years | 2 | 2 | 6 | 7 | 17
  Between 50 and 59 years | 8 | 16 | 27 | 19 | 70
  Between 60 and 69 years | 10 | 12 | 29 | 24 | 75
  >=70 years | 2 | 12 | 13 | 11 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 49 | 32 | 106
  Male | 12 | 27 | 26 | 29 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 3 | 7 | 14
  Not Hispanic or Latino | 19 | 41 | 72 | 54 | 186
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 6 | 8 | 19
  White | 18 | 40 | 67 | 51 | 176
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 42 | 75 | 61 | 200
KRAS mut+ [Count of Participants; unit: Participants]
  No | 16 | 34 | 53 | 43 | 146
  Yes | 6 | 8 | 22 | 18 | 54

OUTCOME MEASURES:

1. Primary Outcome: 8-Week Disease Control Rate (DCR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 8 weeks
Population: 12 participants were inevaluable and 2 participants were not applicable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Erlotinib | Arm 2 - Erlotinib + MK-2206 | Arm 3 - AZD6244 + MK-2206 | Arm 4 - Sorafenib
Number analyzed (Participants) | 19 | 36 | 70 | 61
Participants
  Partial Response | 0 | 0 | 3 | 3
  Stable Disease | 6 | 18 | 34 | 25
  Progressive Disease | 13 | 18 | 33 | 33

2. Secondary Outcome: Median Progression-free Survival
Description: Progression-free survival was estimated by Kaplan-Meier method
Time Frame: From the date of drug start to the earliest sign of disease progression or death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 - Erlotinib | Arm 2 - Erlotinib + MK-2206 | Arm 3 - AZD6244 + MK-2206 | Arm 4 - Sorafenib
Number analyzed (Participants) | 22 | 42 | 75 | 61
months | 1.8 [1.6 to 3.5] | 2.5 [1.9 to 3.5] | 2.2 [1.8 to 3.6] | 2.1 [1.8 to 2.8]

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dose of study medication, up to 3 years
Arm/Group | Arm 1 - Erlotinib | Arm 2 - Erlotinib + MK-2206 | Arm 3 - AZD6244 + MK-2206 | Arm 4 - Sorafenib
All-Cause Mortality (participants affected / at risk) | 19/22 | 36/42 | 65/75 | 51/61
Serious Adverse Events (participants affected / at risk) | 3/22 | 13/42 | 29/75 | 24/61
Other Adverse Events (participants affected / at risk) | 21/22 | 42/42 | 75/75 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Erlotinib (N=22) | Arm 2 - Erlotinib + MK-2206 (N=42) | Arm 3 - AZD6244 + MK-2206 (N=75) | Arm 4 - Sorafenib (N=61)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 3 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 (0) | 4 (5)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 1 (1)
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 | 2 (2) | 0 | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Dyspnea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 7 (11) | 5 (5)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Esophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Fatigue (General disorders) | 0 | 0 | 1 (1) | 0
Fever (General disorders) | 0 | 2 (2) | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 (1) | 1 (1) | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
Investigations - Other, specify (Investigations) | 0 | 0 | 1 (1) | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 (1) | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Lung infection (Infections and infestations) | 1 (1) | 0 | 3 (3) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Multi-organ failure (General disorders) | 1 (1) | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 (1) | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 1 (1)
Pain (General disorders) | 0 | 1 (1) | 1 (1) | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Pancreas infection (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0
Renal colic (Renal and urinary disorders) | 0 | 1 (1) | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2) | 3 (3) | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Skin infection (Infections and infestations) | 0 | 1 (1) | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 0 | 1 (2)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 0 | 1 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 | 0 | 4 (5) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 (1) | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Erlotinib (N=22) | Arm 2 - Erlotinib + MK-2206 (N=42) | Arm 3 - AZD6244 + MK-2206 (N=75) | Arm 4 - Sorafenib (N=61)
Fatigue (General disorders) | 2 | 15 | 31 | 26
Diarrhea (Gastrointestinal disorders) | 8 | 24 | 26 | 16
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 3 | 14 | 29 | 24
Rash Acneiform (Skin and subcutaneous tissue disorders) | 11 | 18 | 29 | 3
Nausea (Gastrointestinal disorders) | 7 | 13 | 25 | 12
Vomiting (Gastrointestinal disorders) | 5 | 10 | 27 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 12 | 13 | 18
Anorexia (Metabolism and nutrition disorders) | 6 | 16 | 9 | 15
Increased AST (Investigations) | 5 | 5 | 29 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 11 | 24 | 4
Oral mucositis (Gastrointestinal disorders) | 3 | 13 | 14 | 10
Increased alkaline phosphatase (Investigations) | 2 | 10 | 17 | 22
Weight loss (Investigations) | 3 | 11 | 2 | 5
Increased ALT (Investigations) | 0 | 5 | 22 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 8 | 5
Other skin and subcutaneous tissue disorders, specify (Skin and subcutaneous tissue disorders) | 3 | 3 | 8 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 8 | 15
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 6 | 6 | 5
Increased blood bilirubin (Investigations) | 5 | 2 | 1 | 9
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 10
Hypertension (Vascular disorders) | 0 | 1 | 2 | 7
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 5 | 3 | 2
Increased creatinine (Investigations) | 0 | 5 | 2 | 8
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT01248247/Prot_SAP_000.pdf